CLINICAL TRIAL: NCT00274001
Title: An Open, Randomised, Multicentre, Comparative Trial, to Evaluate the Benefit of Switching From a PI-based Regimen to a Nevirapine-based Regimen on the Quality of Life, Patient Adherence, Patient's Perception of Fat Redistribution and Metabolic Changes, in HIV+ Patients Suffering From Fat Abnormalities
Brief Title: Quality of Life and Changes in Metabolism of Lipids and Glucose After Switching to a Nevirapine-based Regimen in HIV+ Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1100.1362
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections; Quality of Life
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
The purpose of this trial is to compare the effect of switching to nevirapine (Viramune®)-containing regimen on quality of life of patients with fat abnormalities and virological control whilst receiving a PI-based regimen.

DETAILED DESCRIPTION:
Patients will receive one of the current standard of care regimens for the treatment of HIV infection, i.e. nevirapine (Viramune®) must be administered in conjunction with 2NRTIs, as prescribed by the investigator at the study sites. Patients randomized to the nevirapine (Viramune®)-arm of the study will receive 1x200mg tablet once daily for the first 14 days ("lead in" period) and 1x200 mg tablet twice daily at appropriately spaced intervals subsequently, plus their SOC combination of 2NRTIs as prescribed by the investigators (without changing their prior NRTIs). Patients randomized to continue their standard treatment will receive it as prescribed by the investigators. No dose modification of the study drugs is permitted during the trial. The study drug will be dispensed at randomization and every four weeks thereafter until completion of 48 weeks. After 6 months at least of treatment the switch from PI regimen to NVP regimen will be allowed to all patients included in the PI arm according to patient's willingness. In these patients AST and ALT should be checked at time 0 (switch) and every 2 weeks for 2 months.

Study Hypothesis:

Between treatment comparison of Nevirapine-based regimen versus PI-based regimen will be based on a null hypothesis of no treatment difference. The null hypothesis will be no difference between the two arms at week 24 (month 6th), against the alternative hypothesis that the mean change in physical domain of the QoL will be 10 points score (SD=20) and the difference between triglycerides normalized patients will be 20%.

Comparison(s):

The primary analysis on physical domain of QoL will be performed on the changes between last observation carried forward following the LCOF approach (i.e. visit 6 or in case of premature discontinuation visit 5 or 4) and baseline (visit 2) value using fixed-effects ANCOVA model with center and treatment groups as factors and baseline value and MMA type interaction will be also included in the main model.

ELIGIBILITY:
Main Inclusion criteria:

* Subject suffering with clinically evident fat redistribution including the lipodystrophic syndrome and/or with abnormal values of triglycerides, cholesterol and/or insulin resistance
* Subject on treatment with HAART including PIs for at least 9 months, without therapeutic changes for at least 6 months
* Baseline CD4+ >200 cells/mm3
* HIV-1 RNA levels <200 copies/mL at baseline and during the previous 6 months

Main Exclusion criteria:

* Subject with other serious or chronic disease unrelated to HIV
* Subject with active invasive infections
* Subject with Karnofsky score less than 50
* Prior NNRTs experience
* Documented or suspected acute hepatitis within 30 days prior to baseline visit, irrespective of AST and ALT values that are >5 ULN
* Subject receiving hypolipidemic and/or antidiabetic drugs at study entry
* Subjects with central nervous system disease or pre-existing mental disturbance
* Subjects on methadone chronic treatment at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2001-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life (WHOQoL questionnaire) | up to 48 weeks
Change in triglycerides in plasma | up to 48 weeks

SECONDARY OUTCOMES:
Patients perception of fat redistribution | up to 48 weeks
Adherence to therapy | up to 48 weeks
Changes in metabolism of lipids and glucose | up to 48 weeks
Bone mineral loss | up to 48 weeks
Therapeutic drug levels of antiretrovirals (drug plasma level / IC90) | up to 48 weeks
Concentration of antiretrovirals in semen and vaginal secretions | up to 48 weeks
Viral load | up to 48 weeks
Immunological status | up to 48 weeks
Incidence and intensity of clinical and adverse events | up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI Italy
Locations (23):
- Italy (23):
  - Ospedale Regionale, Ancona
  - Ospedale Santa Maria Annunziata, Antella (fi)
  - Clinica di Malattie Infettive, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi di Biella, Biella
  - Istituto di Malattie Infettive, Bologna
  - Ospedale Civile, Brescia
  - Spedali Civili di Brescia, Brescia
  - Ospedale di Circolo di Busto, Busto Arsizio (va)
  - Ospedale SS. Trinità, Cagliari
  - Azienda Ospedaliera Arcispedale S. Anna, Ferrara
  - Ospedale San Martino, Genova
  - Presidio Ospedaliero "A. Manzoni", Lecco
  - Azienda Ospedaliera Carlo Poma, Mantova
  - Ospedale Luigi Sacco, Milan
  - Fondazione Centro S. Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera "Luigi Sacco", Milan
  - Policlinico Universitario, Modena
  - Ospedale A. Cotugno, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale Civile, Piacenza
  - Ospedale Cisanello, Pisa